CLINICAL TRIAL: NCT03010293
Title: Pressure Ulcer-associated Osteomyelitis: Retrospective Evaluation of a Two-stage Surgical Strategy (Debridement With Vacuum-assisted Closure Therapy and Reconstruction) With Prolonged Antimicrobial Therapy
Brief Title: Pressure Ulcer-associated Osteomyelitis: Evaluation of a Two-stage Surgical Strategy With Prolonged Antimicrobial Therapy
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0391
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Bone Diseases, Infectious
Keywords: Antimicrobial therapy; Debridement; Osteomyelitis; Muscular flap; Pressure ulcer; Treatment failure; Vacuum-assisted closure therapy
MeSH Terms: conditions — Bone Diseases, Infectious; Osteomyelitis; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pressure ulcer represents a frequent clinical condition in patient with spinal cord injury or after prolonged Intensive Care Unit (ICU) stay. Osteomyelitis constitutes a severe complication with a poorly known management, and is associated with a high rate of relapse, leading to a high-burden in hospital bed-days, financial cost, surgical intervention, antibiotic use, morbidity and mortality, and nursing care. In our reference center for bone and joint infection management, the medical and surgical strategies are systematically discussed during pluridisciplinary meetings. Most patients benefit from a two-stage surgical strategy (debridement with initiation of vacuum-assisted closure therapy until reconstruction using muscular flap) with prolonged antimicrobial therapy. In this context, our study aims to evaluate this complex approach and to determine risk factors of treatment failure in order to improve patient management, focusing on optimization of empirical antimicrobial therapy after each surgical stage, delay between the two surgical stage, and duration of antimicrobial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e age ≥ 18 year-old) with a osteomyelitis complication following a pressure ulcer who benefited from a two-stage surgical strategy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pressure ulcer-related osteomyelitis
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Failure of a two-stage surgical strategy in patient with ischiatic or sacral pressure ulcer-associated osteomyelitis | 2 years after antibiotic therapy disruption
  Treatment failure will include: 1) local clinical and/or microbiological relapse; and/or 2) need for additional surgery after surgical reconstruction by muscular flap; and/or 3) death of septic origin.

SECONDARY OUTCOMES:
Risk factor for treatment failure of a two-stage surgical strategy with prolonged antimicrobial therapy in patient with ischiatic or sacral pressure ulcer-associated osteomyelitis | 2 years after antibiotic therapy disruption
  Risk factor for treatment failure will particularly focus on empirical antimicrobial therapy after each surgical stage, delay between the two surgical stage, optimization of local condition (including discharge, colostomy) and duration of antimicrobial therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Principal Investigator — Centre de reference des infections ostéo-articulaires, Hôpital de la Croix-Rousse
Locations (1):
- Centre de référence des Infections Ostéo-articulaires-Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Derived] Triffault-Fillit C, Valour F, Guillo R, Tod M, Goutelle S, Lustig S, Fessy MH, Chidiac C, Ferry T; Lyon BJI Study Group. Prospective Cohort Study of the Tolerability of Prosthetic Joint Infection Empirical Antimicrobial Therapy. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e00163-18. doi: 10.1128/AAC.00163-18. Print 2018 Oct. PMID 30038037
- [Derived] Andrianasolo J, Ferry T, Boucher F, Chateau J, Shipkov H, Daoud F, Braun E, Triffault-Fillit C, Perpoint T, Laurent F, Mojallal AA, Chidiac C, Valour F; Lyon BJI study group. Pressure ulcer-related pelvic osteomyelitis: evaluation of a two-stage surgical strategy (debridement, negative pressure therapy and flap coverage) with prolonged antimicrobial therapy. BMC Infect Dis. 2018 Apr 10;18(1):166. doi: 10.1186/s12879-018-3076-y. PMID 29636030
- See also: Related Info — http://www.crioac-lyon.fr